CLINICAL TRIAL: NCT06222112
Title: Experience Life, Needs and Expectations of Families of Older Polyhandiccaped Persons
Acronym: PolyAge
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM23_0212
Record Dates: First submitted 2024-01-03; First posted 2024-01-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-01

CONDITIONS: Polyhandicap

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general objective of PolyAGE is to explore the life experience of familial caregivers of aging persons with polyhandicap (>= 35 years). The investigators will question parents (objective 1) and siblings (objective 2) about the experiences, the social representations, the needs and the expectations, as well as the mechanisms associated with their choices about their children with polyhandicap. The objective 3 is to co-analyze parents' and siblings' experiences regarding the aging of their relatives with polyhandicap.

DETAILED DESCRIPTION:
Context Polyhandicap as a chronic complex disability condition, lead to a combination of profound intellectual disability and serious motor deficit, resulting in the extreme restriction of autonomy and communication. Due to the improvement of preventive actions and supportive care, the life expectancy of these persons is increased In order to assess the issues associated with the aging of people with polyhandicap (an emerging and underexplored phenomenon), life experiences, social representations, specific needs and expectations of familial caregivers (parents and siblings) need to be explored. It is essential to better understand these phenomenon in order to better support and assist these families. The PolyAGE project relies on an interdisciplinary approach, based on social and human sciences (social psychology of health) and public health. PolyAGE is based on a solid network including engaged and volunteer actors.

Objectives The general objective of PolyAGE is to explore the life experience of familial caregivers of aging persons with polyhandicap (>= 35 years). The investigators will question parents (objective 1) and siblings (objective 2) about the experiences, the social representations, the needs and the expectations, as well as the mechanisms associated with their choices about their children with polyhandicap. The objective 3 is to co-analyze parents' and siblings' experiences regarding the aging of their relatives with polyhandicap.

Methods

PolyAGE relies on the EVAL-PLH cohort, initiated in 2015, including persons with polyhandicap, familial and institutional caregivers. Eight teams are involved in PolyAGE: 2 specialized reeducation centers (Hendaye et San Salvadour), the J. Bost Foundation, the Groupe Polyhandicap France (family association), 3 university teams (CeReSS and LPS of Aix Marseille university and SantESiH of Montpellier university), 1 epidemiology team (AP-HM).The investigators propose a pluri-methodological mixt approach combining quantitative and qualitative approaches in a socio-contextual and comprehensive perspective:

1. Quantitative approach:

   * Evaluations using standardized self-reported questionnaires: quality of life, coping, emotional intelligence, burden.
   * Parents: data already available (EVAL-PLH cohort: 2 evaluation times 20151-6 and 2020-21).
   * Siblings: data to be collected (phone, mail).
2. Qualitative approach:

   * Evaluations based on interviews (parents and siblings; 1 confounding factor: participant's sex);
   * Combination of interviews content and interpretative phenomenological analysis.
3. Methodological triangulation:

   * Crossing and confrontation of quantitative and qualitative findings. Perspectives
   * Improvement of knowledge and identification of the specific needs/expectations of family caregivers of aging persons with polyhandicap.
   * Understanding the underlying reasons behind the choices made by families in terms of support for aging persons with polyhandicap in order to support the transitions related to the joint aging of persons with polyhandicap and their relatives.
   * Better supporting families in the aging transition (health professionals, health-decision makers).

ELIGIBILITY:
Inclusion Criteria:

* Mother or father (>=18 years) of a with severe polyhandicap aged 35 and over at the time of inclusion
* Person (>=18 years) having at least one parent in common with a person with a severe polyhandicap aged 35 and over at the time of inclusion
* Person agreeing to participate after having been informed of the study's objectives and procedures

Exclusion Criteria:

* Parents and siblings whose inclusion criteria concerning the Persons with severe polyhandicap are not fulfilled
* Parents and siblings who refuse to participate

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with severe polyhandicap aged 35 and over. Severe polyhandicap was defined according to the following criteria:
  * presence of a brain lesion that occurred before the age of 3,
  * IQ below 40 or not assessable,
  * motor handicap: para/tetraparesis or hemiparesis,
  * Gross Motor Function Classification System score of III, IV or V,
  * Functional Independence Measure score below 55
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Experiences of parents of aging persons with polyhandicap | 30 minutes to fill in the booklet and about 60 minutes for the interview
  Evaluations using standardized self-reported questionnaire: quality of life and evaluation based on interviews to be conducted during the present study

SECONDARY OUTCOMES:
Experiences of siblings of aging persons with polyhandicap | 30 minutes to fill in the booklet and about 60 minutes for the interview
  Evaluations using standardized self-reported questionnaire: quality of life and evaluations based on interviews to be conducted during the present study
Crossing and confrontation of quantitative and qualitative findings | 2 months
  A cross of quantitative evaluation (questionnaire) and qualitative evaluation (interviews) by methodological triangulation analysis

CONTACTS AND LOCATIONS:
Overall Officials: karine baumstarck, PI, Principal Investigator — Assistance Publique des Hôpitaux de Marseille (AP-HM)
Locations (7):
- France (7):
  - APHP Hôpital Marin de Hendaye, Hendaye
  - AP-HP Hôpitaux San Salvadour, Hyères
  - Fondation John Bost, La Force
  - Assistance Publique Des Hopitaux de Marseille, Marseille
  - Université Aix Marseille, Marseille
  - Université de Montpellier, Montpellier
  - Groupe Polyhandicap France (GPF), Paris